CLINICAL TRIAL: NCT02578654
Title: Interventions to Improve HIV Care Engagement Within 30 Days After Hospital Discharge Among HIV-infected Patients
Brief Title: Interventions to Improve HIV Care Engagement After Hospital Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Thana Khawcharoenporn, Assistant Professor, Thammasat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MTU-EC-IM-2-082/57
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventions (Experimental): Additional HIV care team daily inpatient round and three telephone calls to remind the upcoming clinic appointment. These interventions are specifically added on "routine care" during the post-intervention period. The routine care does not include the additional round and the three telephone calls and is assessed during the pre-intervention period.
  Interventions: Other: Strategies to improve HIV care engagement

INTERVENTIONS:
Other: Strategies to improve HIV care engagement — Additional HIV care team daily inpatient round and three telephone calls to remind the upcoming clinic appointment. These interventions are specifically added on "routine care" during the post-intervention period. The routine care does not include the additional round and the three telephone calls and is assessed during the pre-intervention period.

SUMMARY:
A quasi-experitmental study of the efficacy interventions, including additional HIV care team daily inpatient round and three telephone calls to remind the upcoming clinic appointment, in improving HIV care engagement within 30 days after hospital discharge among HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients hospitalized at Thammasat University Hospital during the study period

Exclusion Criteria:

* The patients who die during admission, are readmitted prior to 30 days after discharge or with incomplete data
* Readmission episodes of the same enrolled patients during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of HIV-infected patients who come to the designated HIV clinic for follow-up within 30 days after hospital discharge divided by the total number of enrolled HIV-infected patients | 30 days

SECONDARY OUTCOMES:
Factors associated with no follow-up withing 30 days after hospital discharge(analyzed in multivariable logistic regression) | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Faculty of Medicine, Thammasat University, Pathum Thani, Changwat Pathum Thani, Thailand

REFERENCES:
- [Derived] Khawcharoenporn T, Damronglerd P, Chunloy K, Sha BE. Enhanced inpatient rounds, appointment reminders, and patient education improved HIV care engagement following hospital discharge. Int J STD AIDS. 2018 Jun;29(7):641-649. doi: 10.1177/0956462417749420. Epub 2018 Feb 5. PMID 29402187